CLINICAL TRIAL: NCT00635791
Title: A Phase I Safety and Tolerability Study of Vorinostat in Combination With Sorafenib in Patients With Advanced Solid Tumors, With Exploration of Two Tumor-type Specific Expanded Cohorts at the Recommended Phase 2 Dose
Brief Title: Phase I Study of Vorinostat and Sorafenib in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0537.cc; NCI-2013-00413 (Other: National Cancer Institute)
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Solid Tumour; Renal Cell Carcinoma; Non Small Cell Lung Carcinoma
Keywords: Malignant Solid Tumour; Renal cell carcinoma; Non small cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib tosylate and vorinostat (Experimental): Patients receive sorafenib tosylate by mouth twice a day on days 1-21 and vorinostat by mouth every day on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sorafenib; Drug: Vorinostat

INTERVENTIONS:
Drug: Sorafenib — Given by mouth
  Other Names: NexAVAR
Drug: Vorinostat — Given by mouth
  Other Names: Zolinza

SUMMARY:
This phase I trial studies the side effects and best dose of giving vorinostat and sorafenib tosylate together in treating patients with kidney or non-small cell lung cancer. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may stop the growth of solid tumors by blocking blood flow to the tumor. Giving vorinostat together with sorafenib tosylate may kill more tumor cells.

DETAILED DESCRIPTION:
The main purpose of this study is to:

* Evaluate the safety of vorinostat in combination with sorafenib.
* Determine the largest dose of vorinostat + sorafenib that can be given safely to humans.
* Determine if vorinostat + sorafenib are effective in stopping tumors from growing or in decreasing their size.
* Study the side effects of vorinostat + sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Parts A: Histologically or cytologically documented solid tumor malignancy or non-Hodgkin's lymphoma (Part B: renal cell carcinoma, Part C: non-small cell lung carcinoma) with clinical evidence of advanced and/or metastatic disease, which is refractory to established forms of therapy or for which no effective therapy exists, or for which sorafenib alone would be considered by the investigator as an appropriate therapy; patients who have refused available standard therapies would also be deemed eligible
* In Part A, evaluable disease by radiology and/or a recognized serum tumor marker is required; in Parts B and C, measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) is required
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Predicted life expectancy ≥ 12 weeks
* Patients may have had prior therapy, providing the following conditions are met:

  * Patients must have recovered from any treatment related toxicities (with the exception of alopecia) to ≤ CTC grade 1 (fatigue, and neurotoxicity at grade 2 are permissible if stable for > 3 months) prior to registration
  * Chemotherapy: A minimum of 5 predicted half-lives of the agent must have elapsed between the end of treatment and registration on to the study; when half-lives are not available the principle of 2 weeks for once daily medications and 3 weeks for agents given less frequently will be adopted, but discussion with the principal investigator is recommended
  * Hormonal therapy: Patients may have had prior anticancer hormonal therapy provided it is discontinued > 4 weeks prior to registration into the study; however, patients with prostate cancer with evidence of progressive disease may continue on therapy which produces medical castration (eg, goserelin or leuprorelin) provided this was commenced at least three months earlier
  * Radiation: Patients may have had prior radiation therapy that has not exceeded 25% of bone marrow reserve provided that they have recovered from the acute, toxic effects of radiotherapy prior to registration; a minimum of 7 days must have elapsed between the end of radiotherapy to non-target lesions and registration into the study (minimum of 28 days for target lesions)
  * Surgery: Previous surgery is permitted provided that wound healing has occurred prior to registration
* Supportive therapy including bisphosphonates is permissible; previous use of myeloid and erythroid growth factor support is permissible, but not within 2 weeks of commencement of study; primary prophylactic use of myeloid and erythroid growth factors is not permitted within the study, but intervention or secondary prophylaxis is permitted if instituted following the documentation of ≥ grade 3 neutropenia or ≥ grade 2 anemia (hemoglobin)
* International Normalized Ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits; patients receiving anticoagulation treatment with an agent such as warfarin or heparin may be allowed to participate; for patients on warfarin, the INR should be measured prior to initiation of sorafenib/vorinostat and monitored at least weekly, or as defined by the local standard of care, until INR is stable; vorinostat and sorafenib have both been reported to elevate INR in those on coumadin derivatives
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 75 x 10^9/L
* Bilirubin ≤ 1.5 x Upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and/or alanine transaminase (ALT) ≤ 2.5 x ULN (ie, ≤ CTC grade 1) or ≤ 5 x Upper limit of normal (UNL) if patient has documented liver metastases (ie, ≤ CTC grade 2)
* Serum creatinine ≤ 1.5 x ULN
* Patient must be accessible for repeat dosing and follow-up
* Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study; women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration
* Patients must provide verbal and written informed consent to participate in the study, including pharmacokinetic sampling

Exclusion Criteria:

* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's ongoing participation in the study
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Concurrent anticancer therapy (with the exception of hormonal therapies as discussed above)
* Pregnant or breast-feeding females (documented methods of birth control are required in those with reproductive potential)
* Symptomatic brain metastases which are not stable, require steroids, or anti-epileptic medication
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs
* History of grade 3 or greater toxicities with vorinostat or sorafenib previously at equivalent daily doses or lower than those planned on being administered within this study
* Exposure to other histone deacetylase (HDAC) inhibitors (e.g. sodium valproate) within 30 days of planned commencement of study drugs, other exposures to HDAC inhibitor and sorafenib in combination
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= Common Toxicity Criteria for Adverse EffectS (CTCAE) grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
* Use of St. John's Wort or rifampin (rifampicin)
* Known or suspected allergy to sorafenib, vorinostat or any planned agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Any clinically significant malabsorption problem
* Clinically significant, in the investigator's opinion, pre-existing cardiac dysfunction or myocardial infarction within 6 months prior to planned commencement of study drugs
* Any other condition, which in the investigator's opinion, would compromise the safety of the patient or the feasibility of completing the study objectives through the use of this patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 21 days
  The primary objective of this study is to determine the MTD for vorinostat in combination with the recommended dose of sorafenib 400 mg when given daily in a 21-day cycle and thereby establish a recommended Phase 2 dose of the combinations when administered daily in patients with advanced solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: David R Camidge, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States